CLINICAL TRIAL: NCT04220905
Title: Large Polyp Study (LPS) III - Endoscopic Resection of Large Colorectal Polyps: An Observational Cohort Study
Brief Title: Endoscopic Resection of Large Colorectal Polyps: An Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Heiko Pohl, Associate Professor of Medicine, Dartmouth College, White River Junction Veterans Affairs Medical Center
Other Study IDs: CPHS 23578
Record Dates: First submitted 2019-12-27; First posted 2020-01-07 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Colonic Polyp; Colonoscopy; Complication; Recurrence; Duodenal Polyp
MeSH Terms: conditions — Colonic Polyps; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol describes a prospective cohort study. It addresses an important challenge in the prevention of colorectal cancer and duodenal cancer: how to safely and effectively remove large polyps.

DETAILED DESCRIPTION:
Over recent years, a number of studies have been published that have highlighted factors associated with improved efficacy and safety of large polyp resection. Almost all of these studies originate from one large Australian cohort. It is unclear, whether the results are generalizable to other populations. It is important to understand if these findings can be duplicated, to further build on the gained knowledge. At the same time the technology of endoscopic resection is evolving.

Established in 2012, the Large Polyp Study group aims to prospectively examine outcomes related to endoscopic large polyp removal. Enrollment of an ongoing randomized trial of 920 patients has just been completed and a second trial is planned. The primary aim of both trials is to understand whether a specific intervention will reduce the risk of adverse events. The added observational study will complement the trials in different ways: It will enroll patients who might not have been eligible for the trials and allow the application of other resection techniques. The observational study will therefore better represent the average patient who undergoes resection of a large polyp. Furthermore, it will add sample size to examine secondary outcomes with greater power.

This is a continuation of NCT01936948 (Safety of Endoscopic Resection of Large Colorectal Polyps: A Randomized Trial) as a observational cohort.

The continuation was approved by the institutional IRB as part of the initial RCT. At this point the investigators document the observational arm as its own study in this registry.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥18 who presents for an upper endoscopy or colonoscopy and who does not have criteria for exclusion
* Patients with a ≥20mm colon polyp
* Patients with a ≥10mm duodenal polyp

Exclusion Criteria:

* Patients who are receiving an emergency endoscopy
* Patients with coagulopathy with an elevated INR ≥1.5, or platelets <50
* Poor bowel preparation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient who is known to have a large colorectal polyp or duodenal polyp and are referred for resection of the polyp.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe complications | Up to 14 days following the procedure.
  Aggregate of all severe adverse events that occur at the time of the procedure or during and up to 14 days of follow-up. Severe adverse events include bleeding, perforation, postpolypectomy syndrome, and clinical events that require an admission to the hospital.
Completeness of polyp resection | During the procedure
  Complete polyp removal is defined as removal of all visible polyp tissue at the end of the EMR, as assessed by the endoscopist.
Polyp recurrence | Up to 5 years (at next scheduled surveillance colonoscopy).
  Presence of biopsy proven neoplastic polyp tissue at the EMR resection site at surveillance endoscopy following complete polyp resection.

SECONDARY OUTCOMES:
Severe bleeding complications | Up to 14 days following the procedure.
  Severe bleeding is defined as the need for hospitalization, transfusion, a repeat endoscopy, surgery, or interventional radiology, up to 14 days following the procedure.
Perforation | Up to 14 days following the procedure.
  Defined as a complete hole, or full-thickness resection of the muscularis propria (Sydney Classification of Deep Mural Injury Type IV)
Postpolypectomy syndrome | Following the procedure up to 14 days.
  Defined as abdominal pain severe enough to warrant an ED visit or hospital admission and presence of leukocytosis and/or required treatment with antibiotics.
Efficacy of submucosal injectate | During the procedure.
  Volume of solution per lesion size (mL/cm2), time of resection.
Intraprocedural bleeding | During the procedure
  Immediate bleeding that requires endoscopic intervention to stop the bleeding (e.g. clip placement or snare tip soft coagulation or coagulation grasper).
Need for colon resection | Up to 3 years following the procedure.
  Patients who require surgery for polyp removal or as a result of complications related to the EMR or follow up procedures.
Technical skill of the endoscopist | During the procedure
  To perform video based assessment of endoscopic resection skills
Cold snare of duodenal adenomas greater than 10 mm | Up to 3 years following baseline procedure
  Safety, efficacy, recurrence of neoplastic polyp at first surveillance endoscopy, serious adverse events
Cold snare of Paris IIa polyps greater than 20 mm | 1 year following baseline procedure
  Safety, efficacy, recurrence, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, MD, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States